CLINICAL TRIAL: NCT05978479
Title: The Effect of Individualized Education Using the Teach-Back Method Based on Roy's Adaptation Model Given to Patients With End-Stage Renal Disease Receiving Hemodialysis Treatment on Treatment Adherence and the Coping Skills
Brief Title: The Effect of Individualized Education Using the Teach-Back Method Treatment on Treatment Adherence and the Coping Skills
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, ELIF ACAR, PhD student internal medicine nursing, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SaglikBilimleriUEACAR0001
Record Dates: First submitted 2023-05-01; First posted 2023-08-07 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-07

CONDITIONS: End Stage Renal Disease on Dialysis
Keywords: Hemodialysis; End-stage renal failure; Treatment adherence; Fluid and dietary restrictions; Teach-Back Method
MeSH Terms: conditions — Kidney Failure, Chronic; Treatment Adherence and Compliance | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Patients in the intervention group (experimental group) will receive a hemodialysis training booklet and face-to-face training using the "Teach Back Method" in three sessions held every other day. The routine care and treatment of the control group will be continued.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Teach-Back Method (Experimental): The intervention group will be trained using the Teach Back Method in 3 sessions on every other day that will last 45-60 minutes. Training topics are hemodialysis treatment, end stage renal failure, fluid and diet restrictions and their importance, medication adherence and its importance and lifestyle rules. At the same time, patients will take education booklets.
  Interventions: Other: Teach-Back Method
- Control group (No Intervention): No intervention will be given to the patients in the control group.

INTERVENTIONS:
Other: Teach-Back Method — No intervention will be given to the patients in the control group.
  Other Names: Control group
  Arms: Teach-Back Method

SUMMARY:
This study was planned to evaluate the effect of individual education given to adult patients with End Stage Renal Disease receiving hemodialysis treatment, using the Roy Adaptation Model-Based Teach Back Method under the guidance of nurses, on their ability to cope with fluid, diet and medication compliance and their adaptation skills.

DETAILED DESCRIPTION:
The study is a randomized, controlled, two-group intervention trial with pretest-posttest design at three centers. The study will enroll adult End Stage Renal Disease patients receiving hemodialysis treatment who meet the inclusion criteria at the three centers where the study is being conducted. Data for the study will be collected using face-to-face interviews, a patient information form, a hemodialysis treatment information form, the End-Stage Renal Disease Adherence Questionnaire, a Coping and Adaptation Processing Scale, and a "Teach Back Method" questionnaire. Patients participating in the study will receive an educational booklet that will be completed after obtaining expert opinion based on the literature from the researcher. Patients in the intervention group will be trained by the researcher using the "Teach Back Method" in three sessions. Each session will last 45-60 minutes. From the 2nd week of the study, patients' questions will be answered and a 15-minute retraining session will be made in every two weeks. Patients in the control group will undergo a pretest and a posttest, and their routine care and treatment will continue. At the end of the study, patients in the control group will take training booklets.

ELIGIBILITY:
Inclusion Criteria:

* Hemodialysis treatment for 4 hours, three times a week for at least 3 months with a diagnosis of end-stage renal failure,
* Individuals between the ages of 18 and 65 years,
* Having no speech, vision or hearing problems,
* Be able to speak, read and write in Turkish,
* Patients who have voluntarily to participate and informed consent form in the study.

Exclusion Criteria:

* Those who do not participate or agree to participate in training,
* The general situation is not suitable for questioning,
* Those diagnosed with a cognitive disease such as dementia.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2023-09-04 (Estimated); Primary Completion 2023-12-08 (Estimated); Study Completion 2023-12-08 (Estimated)

PRIMARY OUTCOMES:
Effect of education conducted with the "Teach Back Method" on treatment adherence | Twelve weeks
  In hemodialysis patients,conditions such as dialysis treatment,medication,fluid and diet intake should be applied in harmony with the patient's life.The effect of educating patients in the intervention group with the "Teach Back Method" on the End-Stage Renal Disease Adherence Questionnaire and treatment adherence is evaluated.The End-Stage Renal Disease Adherence Scale is a scale that evaluates the patients' participation in hemodialysis treatment,their use of medication,their compliance with diet and fluid restriction.The validity and reliability of the scale were based on 9 items.The total score that can be obtained from 6 items varies between 0-1200.As the score obtained from the scale increases,the level of adherence to treatment increases.Compliance with scale hemodialysis treatment;It is a valid and reliable self-report tool that evaluates participation in hemodialysis treatment in all areas,including drug use,compliance with diet and fluid restriction.
The effects of the Teach Back Method education on coping with and adaptation to hemodialysis treatment. | Twelve weeks
  This study evaluates the effect of training received by patients in the intervention group using the "Teach Back Method" with Coping and Adaptation Processing Scale to cope with and adaptate to hemodialysis treatment.
  The scale consists of 47 items and 5 sub-dimensions. Scale sub-dimensions; Solution Finding and Focusing, Physical and Decision Making, Attention Process, Systematizing Process, and Learning and Relationship Building. Scale items are of 4-point Likert type. While calculating the Coping and Adaptation Scale score, it is obtained by summing the numerical values of the answers given for each item (reverse scoring is done for the Physical and Decision Making sub-dimension). The total score that can be obtained from the scale varies between 47-188. An increase in the score obtained from the scale is interpreted as more effective coping methods are used.
The effectiveness of using the Teach Back Method in hemodialysis patients | Ten weeks
  The effectiveness of the training for patients in the intervention group will be evaluated every two weeks using the "Teach Back Method" questionnaire.
  In order to evaluate the knowledge, behaviors and skills acquired by the patients during the follow-ups, the Tell What You Have Learned Questionnaire, prepared by the researcher in line with the literature will be used. The Tell What You Have Learned Questionnaire consists of topics including drug therapy, interdialytic weight gain, diet management, fluid consumption, symptom management and physical activity. The Tell What You Have Learned Questionnaire consists of a total of 18 questions, one for each measuring knowledge, behavior and skill for each subject. Patients are expected to answer correctly at least 75 percent of the questions about knowledge, behavior and skill learning areas.

SECONDARY OUTCOMES:
The Effect of the Training given with the Teach Back Method on Interdialytic Weight | Twelve weeks
  The effect of the individual training given with the teach-back method on the difference between the weight measured before and after dialysis will be examined.
The effect of training given with the Teach-Back Method on the amount of ultrafiltration | Twelve weeks
  The effect of the training given with the teach-back method on the amount of ultrafiltration will be examined.
  The amount of ultrafiltration is an objective measure of how the patient manages and adheres to fluid intake. The amount of ultrafiltration can be defined as the difference between the weight measured after the previous dialysis and the weight measured before the current dialysis application. A high amount of ultrafiltration indicates poor compliance with liquid restrictions. As an indicator of compliance for liquid restriction, it is desirable that the amount of ultrafiltration be between 3-5% of dry weight or below 4-4.5%.
The effect of training given with the Teach Back Method on arterial blood pressure | Twelve weeks
  The effect of training given with the teach-back method on arterial blood pressure will be examined.
The effect of training given with the Teach Back Method on dialysis adequacy (Kt/V) | Twelve weeks
  The effect of individual training given with the teach-back method on dialysis adequacy will be examined.
  Dialysis adequacy; It refers to the dialysis dose measured by solute removal, which includes all functions of the kidney. Adequate dialysis is the dialysis dose in which there are no uremic symptoms, biochemical parameters are within the normal range, and one feels good mentally and psychologically. Dialysis adequacy should be evaluated by clinical evaluation, laboratory findings and kinetic indicators. Kt/V; It is calculated by multiplying the urea clearance of the dialyzer by the dialysis time and dividing by the urea distribution volume. It will be taken from the patient file. The target Kt/V for hemodialysis should be between 1.2 and 1.4.

CONTACTS AND LOCATIONS:
Overall Officials: Elif Acar, Msc., Principal Investigator — University of Health science; Semiha Akın, Prof., Principal Investigator — University of Health science